CLINICAL TRIAL: NCT05049759
Title: Development, Testing and Implementation of a Physical Activity Intervention for Youth With Anxiety and Depression -Confident, Active and Happy Youth
Brief Title: Physical Activity Intervention for Youth With Anxiety and Depression -Confident, Active and Happy Youth
Acronym: CAH-Y
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Strathclyde (Other); Western Norway University of Applied Sciences (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30912
Record Dates: First submitted 2021-08-19; First posted 2021-09-20 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Anxiety; Depression; Physical Activity; Activity Trackers
Keywords: Anxiety; Depression; Physical Activity; Youth
MeSH Terms: conditions — Anxiety Disorders; Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Feasibility trial to establish acceptability and feasibility of the developed intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility testing (Experimental): The feasibility trial, aims to assess the feasibility of the intervention, including assessment of acceptability and outcome measures. Twenty youths with anxiety and/or depressive symptoms will be recruited to the intervention. Physical activity will be measured using the Actigraph GT3X+ monitor at baseline and post-intervention. Outcome measures concerning symptom change will be assessed (anxiety and depression). Semi-structured qualitative interview with participants, caregivers and referring specialists will help identify possible contextual and practical factors associated with delivery of the intervention and explore acceptability of assessment procedures, the intervention, and perceived benefits and barriers to participation.
  Interventions: Behavioral: Confident, Active and Happy Youth

INTERVENTIONS:
Behavioral: Confident, Active and Happy Youth — The three target goals of the intervention (confident, active and happy) link closely to the core symptoms of internalizing disorders. Thus, a core symptom of anxiety is a lack of confidence in one's ability to cope with a given fearful situation. The ensuing behavioral reaction is avoidance of the situation and/or enduring it with excessive discomfort. Similarly, a core symptom of a depressive disorder is lowered mood. Regarding both depression and anxiety, both disorders are associated with less physical activity, and low levels of physical activity conversely help maintain the disorders. As such, the aim is to alleviate symptoms and supplement ongoing treatment in CAMHS.
  Other Names: CAH-Y

SUMMARY:
Prevalence of mental health problems and disorders in children and adolescents (hereafter youths) are estimated at 13.4% of which anxiety and depressive disorders account for more than half of these disorders. These rates are increasing, putting a large strain on child and adolescent mental healthcare services (CAMHS) to provide cost-effective treatments with documented long-term effects. However, even when provided the best evidence based treatment, between 40-50 % do not recover and continue to report significant symptom burdens. Thus, there is an immediate need for supplementary and/or new treatment approaches. Physical activity as a supplementary treatment may be one such approach. However, research investigating this approach within this population is scant. This protocol paper describes the development and feasibility trial of a physical activity based intervention targeting anxiety and depressive symptoms in youth.

The current study will be based on the UK Medical Council Research Framework (MRC) for developing and evaluating complex interventions. The study will initially focus on the first two phases of the MRC framework. In line with phase one of this framework, key intervention components have been identified in preliminary work, which draw on the effects of moderate to vigorous physical activity, inhibitory learning theory and self determination theory. These components are to be developed into an intervention to be used in CAMHS. Twenty youths with anxiety and/or depressive symptoms will be recruited to the intervention. Physical activity will be measured using the Actigraph GT3X+ monitor at baseline and post-intervention. Outcome measures concerning symptom change will be assessed (anxiety and depression). Semi-structured qualitative interview with participants, caregivers and referring specialists will help identify possible contextual and practical factors associated with delivery of the intervention and explore acceptability of assessment procedures, the intervention, and perceived benefits and barriers to participation.

This study will contribute to the development of evidence-based, patient-informed supplementary physical treatment interventions for youth with internalizing disorders in contact with CAMHS. The goal is to examine new avenues of treatment that ultimately may improve upon current treatment outcomes of these disorders.

DETAILED DESCRIPTION:
In order for health authorities to be able to respond to the current high demand on mental health services in youth, current treatment interventions need to be examined. The need for augmented and/or supplementary interventions is pressing. Physical activity appears to be a promising, low-risk intervention that may serve this purpose and provide long-term protective health benefits. Despite the potential gain from including physical activity in CAMHS treatments, to our knowledge, no previous study has examined the use of a physical activity program in CAMHS as a supplementary treatment in youth's with anxiety and/or depression. Furthermore, there is a paucity of studies of high methodologically quality examining this topic.

It is the aim of the current study to address this shortcoming by developing a theoretically based physical activity intervention to supplement existing treatment for youth with internalizing disorders (Confident, Active and Happy Youth: CAH-Y).

The current research and intervention development will be based on the UK Medical Council Research Framework (MRC) for developing and evaluating complex interventions.

The MRC framework strongly recommends carrying out feasibility testing prior to any full-scale trial. In line with this recommendation and phases, one and two of the MRC framework, this study proposes to develop and examine the feasibility of recruitment, retention and acceptability of a physical activity intervention for youth with anxiety and/or depression treated in CAMHS. This work will lay the groundwork for later phases and a definitive RCT.

Methods Development of the intervention The theoretical framework for the CAH-Y intervention will draw on three theories. While not a unified theory, the evidence on the psycho-physiological effect of moderate to vigorous physical activity in regards to mood and anxiety disorders in youth specifically and youth mental health in general, indicates a plethora of causal pathways and positive effects. Primarily modulation of monoamines (e.g., increase in serotonin levels), and HPA axis regulation are assumed to be of importance in relation to anxiety and depression. Secondly, Self Determination Theory is a framework with which to understand participant experiences with physical activity and their motivation towards physical activity. The framework focuses on intervention components that can enhance learning and intrinsic motivation concerning both increased activity and behaviour and symptom change. Regarding motivation, evidence suggests that in order to establish physical activity behaviour change, individuals must be either in the 'preparation' or in the beginnings of an 'action' stage of change. Thus, in order to increase physical activity, it is critical that participants are engaged and ready to change behaviour. The final theoretical foundation is inhibitory learning theory which provides a generic framework to understand the bi-directional interaction between cognition, affects and behaviour in regards to anxiety and depression and in particular the role of (physical activity) avoidance as a contributor to and a maintaining factor in these disorders.

Drawing on evidence from CBT treatment for youths with anxiety disorders, evidence suggests that group treatment is equally as effective as individual treatment in CAMHS populations. Furthermore, group treatment provides a number of benefits compared to individual treatment with the current patient group that render this format superior.

Feasibility testing of the intervention Once the CAH-Y intervention is developed a feasibility, study will be conducted with the goal of investigating intervention feasibility, appropriateness and practicality of the designed intervention in the proposed setting, and appropriateness of the assessments. In addition, as noted in the study aims, an effect size will be estimated for a subsequent randomized controlled trial based on previous literature (MRC - Phase 3). The feasibility study is a single arm, non-randomized pre-post control study.

The CAH-Y intervention will be part of the treatment package available to youth in contact with child and adolescent mental health services (CAMHS), Haukeland University Hospital. The CAH-Y intervention is organized within the CAMHS context and will be delivered by personnel employed in this organization. CAMHS is organized at the same intervention level as ordinary hospital services (Haukeland University Hospital, Bergen, Norway) and is as such a tertiary specialized service. In the Norwegian context, this is the primary source of treatment for youth with mental health disorders.

Study population and eligibility Youth are referred to the treatment program from their attending psychiatrist or psychologist at the local CAMHS.

Recruitment

Youth will be recruited from CAMHS, Department of Child and Adolescent Psychiatry, Haukeland University Hospital, Norway. Given that CAH-Y is organized within CAMHS, this enables easy access to potential participants and streamlined recruitment strategies. In practice, this translates into:

* uncomplicated dispersion of information regarding the intervention to the departments and mental health professionals via intranet, email and/or physical/digital meetings
* ease of implementing an in-house digital referral system
* a low threshold for communication between the CAH-Y team and the referring specialist Consent Written consent is obtained from parents and the children. The regional ethical committee has approved the feasibility study (REK NR. 30912).

Feasibility procedures After referral to CAH-Y and assessment of eligibility, eligible youth and their primary caregivers are invited to attend a recruitment and inclusion interview. This interview will take place in the CAH-Y facilities, and the interview will serve several purposes. In the interview, therapists will provide further information about the intervention and study details, clarifying any questions and/or concerns, obtaining written consent and therapists collect and check the questionnaires included in the invitation for the recruitment interview. Moreover, additional questionnaires will be filled out (see primary and secondary outcome measures section), medical information gathered (height and weight), participants will be provided an Actigraph activity monitor to be worn the next seven days and an activity diary to fill out. In addition, a short qualitative interview exploring participant and caregiver views on physical activity will be conducted. Finally, the youth and caregivers will be given a tour of the CAH-Y facilities in order to familiarize them with the setting.

The next contact with the youth will be the first session of the CAH-Y program, which will be between one to a maximum of three weeks after the recruitment and inclusion interview. At this point, participants will also return the Actigraph monitors and activity diaries. The intervention then progresses bi-weekly the next seven weeks. The day before every session, the participants will receive a SMS reminder of the session, as well as a link to the website explaining the program for this the particular session. This is in order to remind the participants of the session clarify what is expected and encourage participation.

Following the last session of the intervention, participants will receive an invitation to attend a post-intervention interview, one to a maximum of three weeks following last intervention session. In this interview, questionnaires relating to symptom change will be completed, biometric data will be gathered and a short qualitative interview exploring the views of the participant and his/her caregivers in relation to the intervention will be done. At the end of the interview, participants will be provided an Actigraph activity monitor to be worn for the next seven days and a complementing activity diary. After these seven days have elapsed, a research assistant will gather the Actigraph. Independently of this assessment with the participant, a short qualitative interview with the referring specialist will also be conducted by the PI.

At six months post-intervention, the participants and their caregivers will be invited to attend a follow-up interview. In this interview, questionnaires relating to initial symptoms will be filled out anew, and a new short qualitative interview exploring views possible negative and/or positive effects of the intervention will be done. It the end of the interview, participants will be provided an Actigraph activity monitor to be worn for the next seven days and a complementing activity diary. After this time-period, the Actigraph will gathered by a research assistant.

Comparison group In the feasibility study in phase 2, no comparison group will participate. Participants will serve as their own controls. Pre- and post-treatment results will be compared.

Measures Apart from the measures that participants and their caregivers fill out at home, all other measures and assessments will be conducted in the CAH-Y facilities.

Socio-demographic characteristics and psychiatric conditions Feasibility outcomes Participant-centered outcome measures. Timing Measures will be assessed at baseline (pre-intervention interview) and at the latest two weeks after completing the intervention in phase 2. Follow-up outcome will be assessed six months post-intervention.

Sample size As this will be the feasibility study to inform the design of the future definitive RCT, a target sample of 20 youth participants will be recruited for estimation of the intended variables.

Statistics and data analysis Quantitative data will be analyzed using SPSS version 22.0 for Windows.

Quantitative summaries regarding feasibility data will be presented in tables and will include:

* number of potential participants referred
* number of participants assessed eligible, and assessed reason for non-eligibility
* attendance and retention rates Baseline data for participants will also be presented in charts as well as any possible participant missing data (questionnaires and Actigraph). Descriptive data will use 95% confidence intervals (mean and standard deviations). Baseline differences between groups (e.g. age, activity level, BMI, number of mental health disorders and questionnaire outcomes) will be analysed using one-way ANOVA. Nominal data (e.g. gender, ethnicity, social class, participation in school physical activity) will be analysed using Chi-square analyses. However, as mentioned the feasibility study is underpowered to detect any effects reliably. Thus, quantitative feasibility outcomes will be interpreted only as feasibility and pilot data due to lack of statistical power.

Qualitative interviews with participants, caregivers and referring specialists will be analysed utilizing thematic analysis. Accordingly, the written interview data will be reviewed for data familiarization; initial codes will be generated, followed by organizing codes into themes, refining themes, and finally defining themes and sub-themes.

ELIGIBILITY:
Inclusion Criteria:

* Age 8- 17 years
* Symptoms of anxiety and/or depression
* Youth display reduced daily physical activity (less than 30 mins. pr. day and/or does not partake in physical leisure activities, and/or does not participate in physical education in school).
* The youth is motivated to partake in physical activity

Exclusion Criteria:

* Physical activity is not advised for medical reasons
* Severe learning disabilities and the youth is unable to understand the study protocol
* Specific psychiatric disorders including any eating disorder, psychosis
* Severe challenging behavior or other needs requiring constant one to one support

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Objective measure of activity change | Pre-treatment, post-treatment (max. 2 weeks following end of treatment) and six months post treatment (long-term)
  Actigraph measurement of youth activity level
Anxiety symptom change | Pre-treatment, post-treatment (max. 2 weeks following end of treatment) and six months post treatment (long-term)
  Spence Child Anxiety Scale, child and parent version (SCAS-C/P). The measure assesses youth anxiety symptoms. The SCAS-C/P comprises 38 items rated on a 4-point scale (0 = never, 1 = sometimes, 2 = often, 3 = always), with possible a minimum score of 0 and possible a maximum score of 114. High scores indicate higher anxiety levels, and lower scores indicate lower anxiety levels.
Affective symptom change | Pre-treatment, post-treatment (max. 2 weeks following end of treatment) and six months post treatment (long-term)
  Short Mood and Feelings Questionnaire, child and parent version (SMFQ-C/P). The measure assesses youth depressive symptoms. The SMFQ consists of 13 items rated on a 3-point scale (0 = not true, 1 = sometimes true, 2 = true), with possible a minimum score of 0 and possible maximum score of 26.Higher scores indicate greater severity of depressive symptoms.
Recruitment rate (number of youth referred/number of youth assessed as eligible). | Pre-treatment
  These descriptive data provide information concerning the feasibility of the program. Tracking of participant recruitment (number of youth referred/number of youth assessed as eligible), Rates will be presented in percent.
Attendance rate (total number of sessions youth attend) | From start of treatment to end of treatment (7 weeks)
  These descriptive data provide information concerning the feasibility of the program. Attendance to the intervention was measured by counting how many sessions each participant attended and then dividing it by the total number of exercise sessions. Attendance is presented as a percent.
Retention rate (number of sessions youth completed before their last session) | From start of treatment to end of treatment (7 weeks)
  These descriptive data provide information concerning the feasibility of the program. Retention rate is defined as the number of participants who remained in the study, i.e. the number of participants who did not drop out.

SECONDARY OUTCOMES:
Key-process-related outcome e.g how did the participant experience the treatment. | Through study completion, an average of 1 year
  Semi-structured qualitative interview

CONTACTS AND LOCATIONS:
Overall Officials: Arne Kodal, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
Data are relevant for feasibility testing, thus not assessed relevant for IPD.

REFERENCES:
- [Derived] Anker EA, Boe Sture SE, Hystad SW, Kodal A. The effect of physical activity on anxiety symptoms among children and adolescents with mental health disorders: a research brief. Front Psychiatry. 2024 May 13;15:1254050. doi: 10.3389/fpsyt.2024.1254050. eCollection 2024. PMID 38818022
- [Derived] Kodal A, Muirhead F, Reilly JJ, Wergeland GJ, Thorsen PJB, Bovim LP, Elgen IB. Feasibility of a physical activity intervention for children and adolescents with anxiety and depression. Pilot Feasibility Stud. 2024 Mar 5;10(1):49. doi: 10.1186/s40814-024-01466-8. PMID 38443992
- [Derived] Kodal A, Muirhead F, Reilly JJ, Wergeland GJH, Thorsen PJB, Bovim LP, Elgen IB. Development and feasibility testing of a physical activity intervention for youth with anxiety and depression: a study protocol. Pilot Feasibility Stud. 2022 Mar 2;8(1):48. doi: 10.1186/s40814-022-01010-6. PMID 35236419